CLINICAL TRIAL: NCT04794816
Title: What Women Want: Real Time Results for Screening Mammography in the Era of Patient-Experience Driven Care
Brief Title: What Women Want: Real Time Results During Screening Mammography in the Era of Patient-Experience Driven Care
Status: Withdrawn | Type: Observational
Why Stopped: 0 participants
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0980; NCI-2021-01501 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0980 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire administration): Participants complete an online questionnaire over 5 minutes regarding information on patient demographics and preferences for receiving real-time appointment imaging results.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study explores why patients may want to receive real-time imaging results during a screening mammogram appointment at an MD Anderson breast imaging center. Real-time imaging results means women receive the results of the mammogram right away during the same clinic visit. Information from this study may help researchers better understand patient preferences to enhance patient-experience driven care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify factors that may influence a patient's desire to receive real-time imaging results during their screening mammogram appointment at a breast center.

OUTLINE:

Participants complete an online questionnaire over 5 minutes regarding information on patient demographics and preferences for receiving real-time appointment imaging results.

ELIGIBILITY:
Inclusion Criteria:

* All female patients scheduled for a screening mammogram at one of our three MD Anderson Cancer Center (MDACC) Breast Imaging Houston Area Location centers
* Patient >= 30 years of age
* Able to complete an electronic informed consent for the study

Exclusion Criteria:

* Patients not scheduled for a screening mammogram at one of the three imaging facilities

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for a screening mammogram at one of three MD Anderson Breast Imaging Houston Area Locations (League City, Diagnostic Imaging (DI)-West Houston and The Woodlands) between December 15, 2020 and March 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Factors that may influence a patient's desire to receive real-time imaging results during their screening mammogram appointment at a breast center | Up to study completion (estimated 2 years)
  Descriptive analyses will include the characterization of patients and preferences by age, location, patient education level, ethnicity, and patient cancer history.

CONTACTS AND LOCATIONS:
Overall Officials: Megan J Kalambo, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT04794816/ICF_000.pdf